CLINICAL TRIAL: NCT01766882
Title: Fluid-Weight, Volume, Sodium, Blood Pressure Management in Hemodialysis by Limiting Intradialytic and Inter-dialytic Exposure to Sodium and Protocol-based Challenge of Post-dialysis Target Weight: A Pilot and Feasibility Trial
Brief Title: Volume,Sodium and Blood Pressure Management in HD
Acronym: VSBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Rajiv Saran, Associate Professor, Internal Medicine/ Associate Director, Kidney Epidemiology & Cost Center, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00054879
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Renal Failure
Keywords: Hemodialysis; Blood Pressure; Hydration Status; Low-sodium diet
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 1. Lower sodium intervention:
     Dietary sodium restriction of ≤2.0 g/day or ≤85 mmol/day
     Lower dialysate sodium at 137 mmol/L.
  2. Progressive Challenge to Post Dialysis Weight:
  The existing target post-HD weight will be progressively challenged by removing additional fluid in small increments.
  Interventions: Behavioral: Lower sodium intervention; Other: Progressive Challenge to Post Dialysis Weight
- Control (No Intervention): Usual care in addition to Blood pressure monitoring and and Hydration status monitoring

INTERVENTIONS:
Behavioral: Lower sodium intervention — 1. Lower sodium intervention:
  1. Dietary sodium restriction of ≤2.0 g/day or ≤85 mmol/day (approximately >180-200mmol/day in the average American diet). Sodium restriction will be implemented using intensive dietary counseling performed weekly by a registered study dietitian using the motivational interviewing technique.
  2. Lower dialysate sodium at 137 mmol/L, if perchance a different concentration of dialysate is used for the enrolled individual, although this is unlikely in both the UM associated units, where for some time now, dialysate concentration of 137 mmol/L is currently being used as standard practice. Investigators will ensure that this sodium concentration is indeed used for all study participants.
  Arms: Treatment
Other: Progressive Challenge to Post Dialysis Weight — The existing target post-HD weight will be progressively challenged by removing additional fluid in small increments, unless clinical evidence of volume depletion or hypotension precludes this challenge in the intervention arm. To avoid the occurrence of intradialytic hypotension, the ultrafiltration rate shall not exceed15 ml/kg/hour and post dialysis weight will not be reduced by more than 0.5 kg per dialysis session. In some patients, this may warrant prolongation of the treatment time to achieve lowering of target post dialysis weight, and this process of target weight reduction may need to continue up to and through the interim assessment phase (6-8 weeks).
  Arms: Treatment

SUMMARY:
The purpose of this study to conduct a pilot, randomized trial in stable HD patients to evaluate the effect of gradual, step-wise reduction of post-hemodialysis target weight, combined with diligent dietary sodium restriction and reduction in dialysate sodium exposure on hydration/volume status and blood pressure (BP) control.

DETAILED DESCRIPTION:
Fluid-weight management is critical for dialysis patients 1, 2. Previous clinical trials have not comprehensively addressed the application of a strategy combining both sodium restriction and a progressive, but gradual challenge of post dialysis target weight for BP and fluid-weight management in hemodialysis (HD). The investigators postulate that a protocolized, stepwise and gradual challenge of post-hemodialysis target weight when combined with diligent dietary sodium restriction <2000mg sodium/day, will lead to better hydration/volume status and BP control in HD patients. A randomized, two parallel arm trial (n=40) among HD patients is proposed, that compares this comprehensive strategy in one group versus 'usual' HD volume/hydration and BP management in the control group. The two primary outcomes are change in volume/hydration status (assessed by bioelectrical impedance analysis-BIA) and change in BP (pre-dialysis in-center readings, home self-monitored readings as well as 44-hour interdialytic BP). Secondary outcomes include change in target post-dialysis weight, slope of on-line relative plasma volume monitoring (using Crit-line monitors), utilization and change, if any, in antihypertensive regimen, change in interdialytic weight gain, objectively assessed salt-appetite, thirst score, frequency of intradialytic hypotension, cramps and duration of post-dialysis fatigue and recovery, time to achievement of dry weight and laboratory parameters (hemoglobin, albumin, brain natriuretic peptide-BNP, aldosterone and hsCRP). The trial will be 14-weeks in duration and will involve comprehensive assessment of study parameters at baseline, middle and end of the trial. It is anticipated that the trial will lead to the the development of a simple and practical approach for volume and BP control in HD patients that will subsequently need to be studied on a larger scale, i.e., a larger, multicenter study with hard endpoints of death and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Stable adult HD patient (age 18-85 years)
* Usual in-center pre-dialysis systolic blood pressure of ≥130mmHg. For this purpose mean of pre-dialysis sitting blood pressures for the past one month prior to randomization will be applied for evaluation of inclusion criteria.
* Able and willing to adhere to study protocol

Exclusion Criteria:

* Recent acute illness (≤1month)
* Recent hospitalization (≤1month)
* Any psychological condition that could interfere with compliance with study protocol.
* Amputation of both lower limbs (due to interference with electric current for BIA measurement)
* Pacemaker, defibrillator, implantable pump, artificial joint, pins, plates or other types of metal objects in the body (other than dental fillings), if their presence interfere with appropriate measurements. In such patients consideration will be given to only doing the calf-BIA measurements and not the total body, at the discretion of the investigators.
* Use of any investigational product or device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Pregnancy or lactation (pregnancy test will be applied only if the patient is in the reproductive age range).
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Pre-dialysis BP measure at Baseline, 6 Weeks and 12 weeks. ABPM measured at baseline and 12 Weeks. Home BP measure through out the 12week period on non-dialysis days
  Change in blood pressure (pre-dialysis in-center blood pressure readings, ABPM and home BP monitoring)

SECONDARY OUTCOMES:
Post-dialysis Weight | 12weeks
  Change in target post-dialysis weight
Heart Rate | 12 weeks
  Change in heart rate
Plasma Volume | 12 Weeks
  Slope of relative plasma volume monitoring
Medication Use | 12 Weeks
  Change in the utilization of antihypertensive medication ( number of medication and dose)
Interdialytic Weight gain | 12 Weeks
  Change in the mid-week interdialytic weight gain
Intradialytic Hypotension | 12 Weeks
  Frequency of intradialytic hypotension; defined as drop in systolic blood pressure associated with symptoms suggestive of low blood pressure such as lightheadedness, dizziness, sweating, etc., or decrease in intradialytic systolic blood pressure to less than 90 mmHg.
Salt Appetite | Baseline, 6 week and 12 week
  A measure of salt taste impairment and preference
Thirst Score | Baseline, 6 week, 12 weeks
  A measure of general thirst.
Post-dialysis fatigue | Baseline, 6 Weeks & 12 Weeks
  A measure of post-dialysis fatigue and recovery after each treatment session
Routine Labs | Baseline and 12Week
  o Routine labs including CBC, renal panel, hsCRP and brain natriuretic peptide (BNP). Interdialytic urine collection for residual renal function (urea and creatinine clearance) estimation will be made. Blood and urine samples will be archived for later analysis for biomarkers such as asymmetric dimethyl arginine (ADMA), plasma aldosterone, and urinary neutrophil gelatinase-associated lipocalin (NGAL), respectively
True Dry Weight | 12 weeks
  Time to achievement of true 'dry weight' (in the intervention arm only)
Hydration Status | 12 weeks
  Change in hydration status, as measured by BIA, using whole body and segmental techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saran, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University Dialysis Unit, Ann Arbor, Michigan
  - University of Michigan Dialyisis Unit, Livonia, Michigan

REFERENCES:
- [Background] Charra B. Fluid balance, dry weight, and blood pressure in dialysis. Hemodial Int. 2007 Jan;11(1):21-31. doi: 10.1111/j.1542-4758.2007.00148.x. PMID 17257351
- [Background] Nanovic L. Electrolytes and fluid management in hemodialysis and peritoneal dialysis. Nutr Clin Pract. 2005 Apr;20(2):192-201. doi: 10.1177/0115426505020002192. PMID 16207656
- [Background] Aybal Kutlugun A, Erdem Y, Okutucu S, Yorgun H, Atalar E, Arici M. Effects of lowering dialysate sodium on flow-mediated dilatation in patients with chronic kidney disease. Nephrol Dial Transplant. 2011 Nov;26(11):3678-82. doi: 10.1093/ndt/gfr092. Epub 2011 Mar 18. PMID 21421595
- [Background] Munoz Mendoza J, Bayes LY, Sun S, Doss S, Schiller B. Effect of lowering dialysate sodium concentration on interdialytic weight gain and blood pressure in patients undergoing thrice-weekly in-center nocturnal hemodialysis: a quality improvement study. Am J Kidney Dis. 2011 Dec;58(6):956-63. doi: 10.1053/j.ajkd.2011.06.030. Epub 2011 Aug 27. PMID 21875769
- [Background] Manlucu J, Gallo K, Heidenheim PA, Lindsay RM. Lowering postdialysis plasma sodium (conductivity) to increase sodium removal in volume-expanded hemodialysis patients: a pilot study using a biofeedback software system. Am J Kidney Dis. 2010 Jul;56(1):69-76. doi: 10.1053/j.ajkd.2009.12.037. Epub 2010 Mar 19. PMID 20303632
- [Background] Ritz E, Dikow R, Morath C, Schwenger V. Salt--a potential 'uremic toxin'? Blood Purif. 2006;24(1):63-6. doi: 10.1159/000089439. PMID 16361843
- [Background] Maruyama C. Improvement of Threshold-Dosage Salt Sensitivity Strips in Evaluating Reduced Salt Diets. The Japanese Journal of Nutrition and Dietetics 1988;46:211-6.
- [Background] Maruyama C. On Salt Taste Sensitivity of Healthy Patients and Patients with High Blood Pressure (Part 2). The Japanese Journal of Nutrition and Dietetics 1990;48:267-71.
- [Background] Bots CP, Brand HS, Veerman EC, Valentijn-Benz M, Van Amerongen BM, Valentijn RM, Vos PF, Bijlsma JA, Bezemer PD, Ter Wee PM, Amerongen AV. Interdialytic weight gain in patients on hemodialysis is associated with dry mouth and thirst. Kidney Int. 2004 Oct;66(4):1662-8. doi: 10.1111/j.1523-1755.2004.00933.x. PMID 15458464
- [Background] McCarley P. Patient empowerment and motivational interviewing: engaging patients to self-manage their own care. Nephrol Nurs J. 2009 Jul-Aug;36(4):409-13. PMID 19715108
- [Background] Sinha AD, Light RP, Agarwal R. Relative plasma volume monitoring during hemodialysis AIDS the assessment of dry weight. Hypertension. 2010 Feb;55(2):305-11. doi: 10.1161/HYPERTENSIONAHA.109.143974. Epub 2009 Dec 28. PMID 20038754
- [Background] Kurtz TW, Griffin KA, Bidani AK, Davisson RL, Hall JE; Subcommittee of Professional and Public Education of the American Heart Association. Recommendations for blood pressure measurement in humans and experimental animals. Part 2: Blood pressure measurement in experimental animals: a statement for professionals from the subcommittee of professional and public education of the American Heart Association council on high blood pressure research. Hypertension. 2005 Feb;45(2):299-310. doi: 10.1161/01.HYP.0000150857.39919.cb. Epub 2004 Dec 20. PMID 15611363
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Background] Urbina E, Alpert B, Flynn J, Hayman L, Harshfield GA, Jacobson M, Mahoney L, McCrindle B, Mietus-Snyder M, Steinberger J, Daniels S; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee. Ambulatory blood pressure monitoring in children and adolescents: recommendations for standard assessment: a scientific statement from the American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the council on cardiovascular disease in the young and the council for high blood pressure research. Hypertension. 2008 Sep;52(3):433-51. doi: 10.1161/HYPERTENSIONAHA.108.190329. Epub 2008 Aug 4. No abstract available. PMID 18678786
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Ware J, Snow K K, Kosnski M, Gandek B. SF-36 Health Survey: Manual and Interpretation Guide. Boston: Health Institute, 1993.